CLINICAL TRIAL: NCT04170751
Title: Effect of Vasopressin vs Norepinephrine on Pulmonary Oxygenation and Lung Mechanics in Patients With Hypertension Therapy During One-lung Ventilation : Preliminary Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2019-0696
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: lobectomy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Patients enrolled were divided into norepinephrine (group N) and vasopressin (group V) by random random numbers. The ratio of each group should be 1: 1.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients, care givers and outcomes assessors are blinded. The investigator should not be included in the blind because the drug must be rate controlled during investigations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group N (Experimental): In group N, 16 mcg / cc of norepinephrine was infused to patients.
  Interventions: Drug: 16 mcg / cc of norepinephrine(group N)
- group V (Experimental): In group V, 0.4 unit / cc of vasopressin was infused to patients.
  Interventions: Drug: 0.4 unit / cc of vasopressin(group V)

INTERVENTIONS:
Drug: 16 mcg / cc of norepinephrine(group N) — In group N, 16 mcg / cc of norepinephrine was infused through the central catheter. Drug titration should be 0.05 mcg / min / kg for norepinephrine and 2 units / hr for vasopressin, until target blood pressure is reached. Drug infusion rate should not exceed 0.3mcg / min / kg for norepinephrine and 10unit / hr for vasopressin for patient's safety.
  Arms: group N
Drug: 0.4 unit / cc of vasopressin(group V) — In group V, 0.4 unit / cc of vasopressin was infused through the central catheter and the respective doses recorded. Drug titration should be 0.05 mcg / min / kg for norepinephrine and 2 units / hr for vasopressin, until target blood pressure is reached. Drug infusion rate should not exceed 0.3mcg / min / kg for norepinephrine and 10unit / hr for vasopressin for patient's safety.
  Arms: group V

SUMMARY:
Hypotension during anesthesia often occurs because reduced systemic vascular resistance and blocked sympathetic nervous system by anesthetic drugs. In patients who are taking hypertension medication, blood pressure drops are exaggerated by inadequate compensation mechanism due to decrease of blood vessel elasticity and desensitization of baroreceptors. In one-lung ventilation (OLV) during thoracic surgery, persistent perfusion of non-ventilatory lungs can lead to increased intra-pulmonary shunt and hypoxemia. As a compensatory mechanism, the gravitational effect and hypoxic pulmonary vasoconstriction occur. Among these, hypoxic pulmonary vasoconstriction is associated with pulmonary vascular resistance. Norepinephrine and vasopressin, which are commonly used in patients with hypotension, affect systemic and pulmonary vascular resistance. However, no studies have been done on lung oxygenation and pulmonary mechanics of these vasoactive drugs in patients undergoing surgery on one lung. Therefore, the purpose of this study is to investigate the effects of vasoactive drugs, norepinephrine and vasopressin, in patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 40-80 years who are planning to have thoracoscopic single lobectomy with unilateral lung ventilation during surgery.
2. Patients taking hypertension drug CCB(calcium channel blocker), ARB(angiotensin II receptor blocker), ACEi(ACE inhibitor, angiotensin converting enzyme inhibitor) at least 4 weeks.
3. American Society of Anesthesiologists (ASA) classification 2~3

Exclusion Criteria:

1. patients with heart failure (NYHA class III~IV)
2. patients who are having moderate obstructive lung disease or restrictive lung disease
3. Low DLCO (< 75%)
4. patients with pulmonary hypertension (mean PAP>25mmHg)
5. patients with liver disease (AST level ≥100 IU/mL or ALT ≥ level 50 IU/L) or kidney disease (Creatine level ≥ 1.5 mg/dL)
6. body mass index (BMI) > 30 kg/m2
7. patients who cannot read explanation and consent form
8. patients who are pregnant

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | about 20 minutes after reaching to the target blood pressure (T2)
  (arterial oxygen partial pressure / fractional inspired oxygen) at the time of T2

SECONDARY OUTCOMES:
lung mechanics: lung compliance | about 20 minutes after reaching to the target blood pressure (T2)
  Compliance= tidal volume/plateau airway pressure (ml/mmHg)
lung mechanics: dead space | about 20 minutes after reaching to the target blood pressure (T2)
  dead space = [(PaCO2 - PetCO2)/PaCO2] * Tidal volume (ml)
lung mechanics: airway pressure | about 20 minutes after reaching to the target blood pressure (T2)
  airway pressure at T2 (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No